CLINICAL TRIAL: NCT05164744
Title: Cardiac Magnetic Resonance for Tissue Characterization-Based Risk Stratification of Cardiopulmonary Symptoms, Effort Tolerance, and Prognosis Among COVID-19 Survivors
Brief Title: Cardiac Magnetic Resonance Tissue Characterization in COVID-19 Survivors
Status: Recruiting | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 21-02023362; R01HL159055-01 (NIH)
Record Dates: First submitted 2021-12-20; First posted 2021-12-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: COVID-19 Pneumonia; COVID-19; COVID-19 Respiratory Infection; COVID-19 Acute Respiratory Distress Syndrome; COVID-19 Lower Respiratory Infection; COVID-19 Acute Bronchitis; Coronavirus Disease 2019
Keywords: coronavirus disease 2019,
MeSH Terms: conditions — COVID-19 | interventions — Echocardiography; Walk Test; Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples will be collected (30-50mL) to examine biomarkers which will be collected by venesection into citrate or anti-coagulated tubes, and comprised of the following: troponin, ferritin, C reactive protein, D dimer, white blood count, hematocrit, hepatic transaminases, erythrocyte sedimentation rate. In addition, blood samples will be partitioned via differential centrifugation, frozen (-80C) and stored for future research (informed by the current protocol) to further test emerging hematological markers reflective of cardiac injury.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnosed with COVID-19: Participants in the study cohort will have been diagnosed with COVID-19 by a PCR (polymerase chain reaction) positive test
  Interventions: Diagnostic Test: Cardiac MRI; Diagnostic Test: Echocardiogram; Diagnostic Test: 6-minute walk test; Diagnostic Test: Questionnaire

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — Patients participate in an NIH funded cardiac MRI to assess their symptoms.
Diagnostic Test: Echocardiogram — Patients participate in an NIH funded cardiac echocardiogram to assess their symptoms.
Diagnostic Test: 6-minute walk test — Patients participate in a 6-minute walk test to assess their symptoms.
Diagnostic Test: Questionnaire — Patients answer a survey-based questionnaire to assess their symptoms.

SUMMARY:
The purpose of this study is to test if visualizing the heart with cardiac MRI/echo will be important in the understanding cardiac function and prediction of cardiopulmonary symptoms, physical effort tolerance, and outcomes in COVID-19 survivors. If successful, the research will allow us to identify the causes of lasting cardiopulmonary symptoms and begin developing cardiac and lung directed therapies accordingly.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is an ongoing global pandemic. Despite substantial short term mortality risk, the overwhelming majority of infected patients survive acute illness, resulting in a growing population at risk for long term events. Cardiopulmonary symptoms are common after COVID-19, as shown by survey data reporting fatigue (53%), dyspnea (43%), and worsened quality of life (44%) 60 days after acute infection, but mechanism and time course of symptoms are unknown. Recent studies and the investigator's preliminary data have shown myocardial tissue abnormalities on cardiac magnetic resonance (CMR) to be common in COVID-19 survivors - raising the possibility that symptoms stem from viral effects on the heart. However, CMR findings to date are limited by small size and clinical data susceptible to referral bias, raising uncertainty as to generalizability. It is also unknown whether altered myocardial tissue properties (fibrosis, edema) impact clinical outcomes.

The central hypothesis of the research is that CMR tissue characterization will be incremental to clinical assessment and cardiac contractile function for prediction of long-term cardiopulmonary symptoms, effort tolerance, and prognosis among COVID-19 survivors. To test this, the investigators will study patients from an active multiethnic New York City registry of COVID-19 survivors: the investigators have already leveraged echocardiographic imaging data from this registry to show that (1) adverse cardiac remodeling (dilation, dysfunction) markedly augments short term mortality, (2) COVID-19 acutely alters left and right ventricular remodeling, and (3) many patients who survive initial hospitalization for COVID-19 have adverse cardiac remodeling - including 40% with left ventricular (LV) dysfunction and 32% with adverse RV remodeling (dilation, dysfunction): the investigator's current proposal will extend logically on the preliminary data to test whether CMR tissue characterization provides incremental predictive utility with respect to reverse remodeling and prognosis. At least 510 COVID-19 survivors will be studied. Echo will be analyzed at time of and following COVID-19 for longitudinal remodeling, as will CMR at pre-specified (6-12, 36 month) follow-up timepoints. Established and novel CMR technologies will be employed, including assessment of cardiac and lung injury, high resolution (3D) myocardial tissue characterization, and cardiopulmonary blood oxygenation. In parallel, QOL, effort tolerance (6-minute walk test), biomarkers, and rigorous follow-up will be obtained to discern clinical implications and relative utility of imaging findings. Aim 1 will identify determinants of impaired quality of life and effort intolerance among COVID-19 survivors. Aim 2 will test whether myocardial tissue injury on CMR is associated with impaired contractility, and whether fibrosis predicts contractile recovery. Aim 3 will determine whether myocardial tissue injury is independently associated with adverse prognosis (new onset clinical heart failure, hospitalization, mortality). Results will address key knowledge gaps regarding COVID-19 effects on the heart necessary to guide surveillance, risk stratification, and targeted therapies for millions of COVID-19 survivors at risk for myocardial injury, cardiopulmonary symptoms, and adverse prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Emergency room presentation and/or hospitalization with COVID-19 infection defined in accordance with established criteria as follows: SAR-CoV2 RT-PCR+ (severe acute respiratory syndrome coronavirus 2 reverse transcription polymerase chain reaction) and at least one of the following symptoms: dyspnea, cough, dysphagia, rhinorrhea, diarrhea, nausea/vomiting, myalgias, fever, syncope/presyncope.

Exclusion criteria:

* Contraindication to CMR (i.e. non-compatible pacemaker/defibrillator) or gadolinium (known hypersensitivity, eGFR (estimated globular filtration rate) <30 ml/min/1.73m2).
* Inability to provide informed consent (e.g. cognitive impairment).
* Unrelated condition (e.g. neoplasm) with life expectancy <12 months prohibiting follow-up.
* Patients with contraindications to gadolinium (known or suspected hypersensitivity, glomerular filtration rate < 30 ml/min/1.73m2) will undergo non-contrast MRI but will not be excluded from this study.
* Patients with known or suspected pregnancy based on Weill Cornell Radiology intake surveys (reviewed by a clinical RN (registered nurse), as well as research personnel) will be excluded from the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study Population will be comprised of 510 patients (Men and women ≥ 18 years old) with documented (SARS-CoV-2 RT-PCR+) COVID-19 infection, inclusive of patients with residual cardiopulmonary symptoms (shortness of breath, fatigue, chest pain) and asymptomatic patients.
Sampling Method: Non-Probability Sample
Enrollment: 510 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Participants with focal fibrosis based on cardiac imaging (MRI and echocardiogram) > 3 months post-COVID-19 (coronavirus disease 2019) diagnosis, at first study visit | Day of first study visit, > 3 months post acute COVID-19 infection
  Focal fibrosis scored on LGE(late gadolinium enhancement) CMR in affected LV segment based on transmural extent of hyperenhanced myocardium at > 3 months post-COVID-19 diagnosis. Further categorized in accordance with established criteria (ischemic: subendocardial or transmural, non-ischemic: mid or epicardial). Total size (% LV myocardium) measured based on segmental scores, further quantified using the full-width half maximum method.
Participants with focal fibrosis based on cardiac imaging (MRI and echocardiogram) at 12-36 months post first study visit | 12-36 months post first study visit
  Focal fibrosis scored on LGE-CMR in affected LV segment based on transmural extent of hyperenhanced myocardium at 12-36 months post first study visit. Further categorized in accordance with established criteria (ischemic: subendocardial or transmural, non-ischemic: mid or epicardial). Total size (% LV myocardium) measured based on segmental scores, further quantified using the full-width half maximum method.
Blood oxygenation of participants at > 3 months post-COVID-19 diagnosis, first study visit | Day of first study visit, > 3 months post- acute COVID-19 infection
  Blood oxygenation in both the heart (LV/RV) and pulmonary arteries measured on QSM (quantitative susceptibility mapping) at > 3 months post-COVID-19 diagnosis, first study visit: conversion from susceptibility to blood oxygenation. Compute left-right heart oxygen saturation difference (ΔSO2) for which venous saturation will be measured in the RV outflow tract/pulmonary artery (PA) junction (analogous to invasive cath), left and right pulmonary artery differential saturation and relative saturation (in relation to the RV), and mixed venous oxygen saturation (SvO2), which will be calculated by subtracting ΔSO2 (on QSM) from arterial oxygen saturation measured by pulse oximetry (obtained at conclusion of CMR exam).
Blood oxygenation of participants at 12-36 months post first study visit | 12-36 months post first study visit
  Blood oxygenation in both the heart (LV/RV) and pulmonary arteries measured on QSM (quantitative susceptibility mapping) at 12-36 months post first study visit: conversion from susceptibility to blood oxygenation. Compute left-right heart oxygen saturation difference (ΔSO2) for which venous saturation will be measured in the RV outflow tract/pulmonary artery (PA) junction (analogous to invasive cath), left and right pulmonary artery differential saturation and relative saturation (in relation to the RV), and mixed venous oxygen saturation (SvO2), which will be calculated by subtracting ΔSO2 (on QSM) from arterial oxygen saturation measured by pulse oximetry (obtained at conclusion of CMR exam).
Lung abnormalities in participants at > 3 months post-COVID-19 infection | Day of first study visit, > 3 months post- acute COVID-19 infection
  Lung abnormalities at > 3 months post-COVID-19 infection graded on high resolution 3D MRA (magnetic resonance angiography) as (1) consolidative or ground glass signal abnormality or (2) linear areas of scarring and fibrosis. A validated semi-quantitative scoring system is then be applied as follows: each of the 5 lung lobes scored based on extent of anatomic involvement where 0=no involvement: 1=<5% involvement; 2=5-25% involvement; 3=26-59% involvement; 4=51-75% involvement; and 5=>75% involvement. The resulting global score is the sum of each individual lobar score (range 0-25).
Lung abnormalities in participants at 12-36 months post first study visit | 12-36 months post first study visit
  Lung abnormalities at 12-36 months post first study visit graded on high resolution 3D MRA (magnetic resonance angiography) as (1) consolidative or ground glass signal abnormality or (2) linear areas of scarring and fibrosis. A validated semi-quantitative scoring system is then be applied as follows: each of the 5 lung lobes scored based on extent of anatomic involvement where 0=no involvement: 1=<5% involvement; 2=5-25% involvement; 3=26-59% involvement; 4=51-75% involvement; and 5=>75% involvement. The resulting global score is the sum of each individual lobar score (range 0-25).
Quality of life (QOL) in participants at > 3 months post-COVID-19 diagnosis, at first study visit based on clinical indices and symptoms assessed by the (Patient-Reported Outcomes Measurement Information System) PROMIS-29 questionnaire. | Day of first study visit, > 3 months post- acute COVID-19 infection
  QOL at > 3 months post-COVID-19 diagnosis evaluated based on scores from the (Patient-Reported Outcomes Measurement Information System) PROMIS-29 questionnaire (0-10 scale per 7 categories) which is represented by a standardized T-score (mean=50, Standard Deviation=10). QOL data will be analyzed as a continuous variable.
Quality of life (QOL) in participants at 12-36 months post first study visit based on clinical indices and symptoms assessed by the (Patient-Reported Outcomes Measurement Information System) PROMIS-29 questionnaire. | 12-36 months post first study visit
  QOL at 12-36 months post first study visit evaluated based on scores from the (Patient-Reported Outcomes Measurement Information System) PROMIS-29 questionnaire (0-10 scale per 7 categories) which is represented by a standardized T-score (mean=50, Standard Deviation=10). QOL data will be analyzed as a continuous variable.
Effort tolerance as measured by a 6-minute walk test at > 3 months post-COVID-19 diagnosis, at first study visit | Day of first study visit, > 3 months post- acute COVID-19 infection
  Effort tolerance > 3 months post-COVID-19 diagnosis quantified via 6-minute walk test, measured as a continuous variable based on total duration walked (during 6-minute test time, or time of patient requested test termination), as well as a age and gender based binary cutoffs employed in prior literature.
  Impaired effort tolerance will be tested both as a binary (<85% predicted) and continuous variable (distance) for statistical analysis.
Effort tolerance as measured by a 6-minute walk test at 12-36 months post first study visit | 12-36 months post first study visit
  Effort tolerance at 12-36 months post first study visit quantified via 6-minute walk test, measured as a continuous variable based on total duration walked (during 6-minute test time, or time of patient requested test termination), as well as a age and gender based binary cutoffs employed in prior literature.
  Impaired effort tolerance will be tested both as a binary (<85% predicted) and continuous variable (distance) for statistical analysis.
Participants with edema based on cardiac imaging (MRI and echocardiogram) at > 3 months post-COVID-19 diagnosis, at first study visit | Day of first study visit, > 3 months post- acute COVID-19 infection
  Edema at > 3 months post-COVID-19 diagnosis: Identified on T2 mapping assessed on a segmental basis corresponding to LGE-CMR. Elevated T2 (i.e. edema) will defined in accordance with established criteria. Myocardial T2 relaxation times extracted from T2 maps after contouring of endocardial and epicardial borders, T2 maps will be analyzed using a 16 segment AHA (American Heart Association) model. T2 values above an established threshold will be indicate presence or absence of edema where T2 value of >80 ms will be used to distinguish edema from healthy myocardium. Global edema assessed as sum of number of affected LV segments. Exploratory analyses test additional indices of edema severity, as assessed based on maximal and mean T2 in all LV segments.
Participants with edema based on cardiac imaging (MRI and echocardiogram) at 12-36 months post first study visit | 12-36 months post first study visit
  Edema at 12-36 months post first study visit : Identified on T2 mapping assessed on a segmental basis corresponding to LGE-CMR. Elevated T2 (i.e. edema) will defined in accordance with established criteria. Myocardial T2 relaxation times extracted from T2 maps after contouring of endocardial and epicardial borders, T2 maps will be analyzed using a 16 segment AHA (American Heart Association) model. T2 values above an established threshold will be indicate presence or absence of edema where T2 value of >80 ms will be used to distinguish edema from healthy myocardium. Global edema assessed as sum of number of affected LV segments. Exploratory analyses test additional indices of edema severity, as assessed based on maximal and mean T2 in all LV segments.
Participants with diffuse fibrosis based on cardiac imaging (MRI and echocardiogram) at > 3 months post-COVID-19 diagnosis, at first study visit | Day of first study visit, > 3 months post- acute COVID-19 infection
  Diffuse fibrosis at 6-12 months post-COVID-19 diagnosis assessed based on extracellular volume (ECV) measured by T1 values in co-registered regions on pre- and post-contrast Modified Look-Locker Inversion (MOLLI): ECV will be calculated via an established formula ECV = (1-hematocrit) * [(1/T1myo post - 1/T1myo pre) / (1/T1blood post - 1/T1bloodpre)].
Participants with diffuse fibrosis based on cardiac imaging (MRI and echocardiogram) at 12-36 months post first study visit | 12-36 months post first study visit
  Diffuse fibrosis at 12-36 months post first study visit assessed based on extracellular volume (ECV) measured by T1 values in co-registered regions on pre- and post-contrast Modified Look-Locker Inversion (MOLLI): ECV will be calculated via an established formula ECV = (1-hematocrit) * [(1/T1myo post - 1/T1myo pre) / (1/T1blood post - 1/T1bloodpre)].
Quality of life (QOL) in participants at > 3 months post-COVID-19 diagnosis, at first study visit based on clinical indices and symptoms assessed by the Minnesota Living with Heart Failure Questionnaire (MLHFQ) | Day of first study visit, > 3 months post- acute COVID-19 infection
  The Minnesota Living with Heart Failure (MLHFQ) scores at > 3 months post-COVID-19 diagnosis range from 0-105 where a higher score indicates more significant impairment in health related quality of life. QOL data will be analyzed as a continuous variable.
Quality of life (QOL) in participants based on clinical indices and symptoms assessed by the Seattle Angina (SAQ) questionnaire at 12-36 months post first study visit | 12-36 months post first study visit
  Seattle Angina (SAQ) questionnaires scored at 12-36 months post first study visit between 0-100 where higher scores indicate better functional status. QOL data will be analyzed as a continuous variable.

CONTACTS AND LOCATIONS:
Overall Officials: Jiwon Kim, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - New York Presbyterian-Brooklyn Methodist Hospital, Brooklyn, New York
  - New York Presbyterian Queens, New York, New York
  - Weill Cornell Medicine/New-York Presbyterian Hospital, New York, New York